CLINICAL TRIAL: NCT03862365
Title: Exploring the Genetics of Neuropathic Pain
Acronym: GeNeup
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Oxford (Other); Danish Pain Research Center (Other); Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Kristian Bernhard Nilsen, Senior Consultant, phd, Oslo University Hospital
Other Study IDs: 2017/1593
Record Dates: First submitted 2018-12-11; First posted 2019-03-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neuropathic Pain; Genetic Predisposition; Polyneuropathies
Keywords: reliability; validity
MeSH Terms: conditions — Neuralgia; Genetic Predisposition to Disease; Polyneuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Whole blood + blood for Expression analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Polyneuropathy with pain: Clinical and diagnostic test evaluation for the establishment of polyneuropathy with pain.
  Interventions: Genetic: Nerve conduction Studies
- Polyneuropathy without pain: Clinical and diagnostic test evaluation for the establishment of polyneuropathy without pain.
  Interventions: Genetic: Nerve conduction Studies
- Diabetic polyneuropathy with pain: Clinical and diagnostic test evaluation for the establishment of diabetic polyneuropathy with pain.
  Interventions: Genetic: Nerve conduction Studies
- Diabetic polyneuropathy without pain: Clinical and diagnostic test evaluation for the establishment of diabetic polyneuropathy without pain.
  Interventions: Genetic: Nerve conduction Studies
- Carpal tunnel syndrome with pain: Clinical and diagnostic test evaluation for the establishment of carpal tunnel syndrome with pain.
  Interventions: Genetic: Nerve conduction Studies
- Carpal tunnel syndrome without pain: Clinical and diagnostic test evaluation for the establishment of carpal tunnel syndrome without pain.
  Interventions: Genetic: Nerve conduction Studies

INTERVENTIONS:
Genetic: Nerve conduction Studies — Patients will be genotyped for comparison of patients With and without pain, With different clinical subgroups as mentioned.
  Other Names: Genetical analysis

SUMMARY:
In the present study the investigators will search for new genetic variants relevant for the development of neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain is defined as "pain caused by a lesion or disease of the somatosensory nervous system". Neuropathic pain is a huge health problem worldwide, with an estimated prevalence of 7-8 % in the general population. In the present study the investigators will search for new genetic variants relevant for the development of this type of pain.

Peripheral nerve lesions only progress to neuropathic pain in some patients, yet is not completely understood why or how. Genetic studies of patients with rare neuropathic disorders have been important for elucidating novel molecular mechanisms of neuropathic pain, and new drugs for neuropathic pain are now being developed based on these findings. By using genetic association studies, one may identify new genetic variants which may help to identify key molecular mechanisms for a larger group of patients with neuropathic pain.

This project will use existing population-based cohorts, as well as establish a specific registry and biobank for patients with neuropathy in order to address these specific needs. This will allow the investigators to identify a large number of individuals with probable neuropathic pain and individuals with pain-free peripheral neuropathy (disease controls). International collaboration will contribute to study a large group of patients, which will be important in order to reach the project's goals. The results from the project are expected to increase current knowledge on the mechanisms of neuropathic pain, opening up new opportunities for innovative and improved treatments.

Dissemination of results will be organized in close collaboration with patient representatives, and will be done regularly throughout the course of the project. The will focus both on internal dissemination to the participating hospitals, and external dissemination through participation in conferences, submissions to scientific journals and by publishing patient-friendly information booklets and proactively informing media outlets and patient organizations.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is between 18 and 70 years old.
2. The patient has consented.
3. The patient is referred for evaluation of possible distal symmetric polyneuropathy (DSPN).
4. The patient has filled out the questionnaires.

Exclusion Criteria:

1. The patient is too sick to participate (eg. bedridden, fever).
2. The patient is unable to consent (eg. dementia, speech problems, psychiatric disorder).
3. Inflammatory acute polyneuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are referred for suspected distal symmetric polyneuropathy and meet the inclusion criteria, will be included in the project. Furthermore, there will be collected blood tests from patients with definite and probable polyneuropathy.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic variants associated with neuropathic pain. | Baseline
  Relevant genotypes will be found using genome-wide association study (GWAS) methodology, ie. with no assumptions regarding which genetic variants that may be relevant (no hypotheses regarding specific variants). This is going to be conducted by using array genotyping (SNPs) in order to identify genetic variants that might be associated with neuropathic pain. Genetic variants will be defined and named according to standard practice, without any room for local or study specific adaptations.
Phenotype; neuropathic pain yes/no | Baseline
  Patients will be divided in two groups; neuropathy With pain (= neuropathic pain) and neuropathy without pain. For definition of neuropathic pain, the Neupsig guidelines (Finnerup et al, Pain 2016) will be used.It is estimated that about 600 patients will be included yearly for this purpose
Phenotype; subgroup analysis of patients with neuropathic pain based on grading of pain | Baseline
  Patients with neuropathic pain will be further subdivided in groups based on pain reports. Pain will be graded using validated questionnaires. The "Brief Pain Inventory-BPI" (Cleeland et al, 1994) questionnaire will be used as primary resource for pain grading, on a scale from 0 to 10 (0: no pain, 1-3: mild pain, 4-10: strong pain).

CONTACTS AND LOCATIONS:
Overall Officials: John Anker Zwart, M.D., Study Chair — Oslo University Hospital; David Benett, M.D., Principal Investigator — University of Oxford; Ina Hjelland, M.D., Principal Investigator — Haukeland University Hospital; Margreth Grotle, Pr., Principal Investigator — Oslo Metropolitan University; Marie Bu Kvaløy, M.D., Principal Investigator — Helse Stavanger HF; Trond Sand, M.D., Principal Investigator — St. Olavs Hospital; Sissel Løseth, M.D., Principal Investigator — University of North Norway; Troels Jensen, M.D., Principal Investigator — Danish pain research senter
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Helse Stavanger HF, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spildrejorde M, Dunker O, Allen SM, Kvaloy MB, Uglem M, Hjelland I, Loseth S, Bennett DL, Zwart JA, Winsvold BS, Gervin K, Selmer KK, Nilsen KB. Genome-wide association study of neuropathic pain. Pain. 2025 Nov 21. doi: 10.1097/j.pain.0000000000003848. Online ahead of print. PMID 41359007